CLINICAL TRIAL: NCT00239096
Title: Losartan in the Prevention of Sodium Retention and Ascites in Liver Cirrhosis - a Prospective Randomized Long-Term Study
Brief Title: Prevention of Decompensation in Liver Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Lundbeck Foundation (Other); University of Southern Denmark (Other); Else Poulsen Mindelegat (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VF20040245; Eudra CT: 2005-001191-12
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2005-10-14 (Estimated); Status verified 2005-10

CONDITIONS: Alcoholic Liver Cirrhosis; Ascites
Keywords: alcoholic liver cirrhosis; ascites; sodium retention
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Ascites; Hypernatremia | interventions — Losartan; Pharmaceutical Preparations

INTERVENTIONS:
Drug: losartan (drug)

SUMMARY:
The purpose of this study is to determine whether losartan, an angiotensin II blocker prevents the sodium retention in patients with liver cirrhosis and by that reduces the fluid retention. Moreover is the purpose to asses whether losartan is antifibrotic.

DETAILED DESCRIPTION:
Patients with cirrhosis tend to retain sodium and water leading to the development of ascites, which in the terminal stage of decompensation cannot be eliminated despite the use of massive diuretic treatment. These decompensated patients have a very high mortality of 50 % within 3 years and morbidity, and until now no symptomatic treatment has been able to improve the prognosis.

It has been hypothesized that ascites and edema develop first due to renal sodium retention secondary to increased activity of hormones like angiotensin II and aldosterone, which may be stimulated by reduced arterial filling caused by systemic vasodilatation, and secondly due to liver fibrosis which may cause lymphatic overflow and formation of ascites.

Decreased central volume filling is believed to stimulate baroreceptors with activation of the renin-angiotensin-aldosterone system, the sympathetic nervous system and arginine vasopressin .

In cirrhotic patients systemic vasodilatation with hypotension, tachycardia, increased cardiac output and increased plasma volume has been thought to be caused by increased levels of vasodilating substances like nitric oxide (NO), but blocking NO synthesis using N(G)-monomethyl-L-arginine-acetate (L-NMMA) did not favorably influence renal sodium excretion, probably due to an important role of NOS in renal sodium handling .

It is evident that the pathophysiology of the development of excessive sodium and water retention in cirrhotic patients is insufficiently elucidated, and that an increased knowledge in this field may improve the therapeutic possibilities. Patients with cirrhosis without ascites have normal or increased glomerular filtration rate (GFR) and normal or suppressed plasma levels of renin, angiotensin II and aldosterone. Later renal blood flow and GFR may be decreased and patients have avid tubular sodium reabsorption as they can produce a virtually sodium-free urine. These functional renal changes regress after transplantation with a normal liver. Suggestions have been made that overfilling rather than central underfilling precede ascites formation. In any case blocking the mineralocorticoid receptor with spironolactone is an effective diuretic treatment in many cirrhotic patients, and this points to the importance of the distal part of the nephron in the mediation of excess sodium reabsorption.

Angiotensin II (ANG II) binds to the AT1 receptor localized to renal glomeruli and tubules, the adrenals and arterioles, not only efferent arterioles in the kidneys, but also resistance vessels of the systemic vasculature. In the adrenals ANG II stimulates aldosterone secretion. In addition it has been shown in rats that the expression of the vasopressin receptor V2 is upregulated by ang II, an effect expected to increase water reabsorption (10). Most likely ANG II aggravates the portal hypertension due to stimulation of stellate myofibroblasts, and this may be part of the circulus vitiosus which should be broken in cirrrhosis. In another volume retaining disorder - heart failure - blockade of the renin angiotensin aldosterone system has been shown to be extremely effective in retarding progression of the disease.

Treatment of cirrhotic patients with ACE-inhibitors has been tried but was poorly tolerated since blood pressure and GFR decreased. In one study, however, the addition of a low dose of Captopril to furosemide and spironolactone increased natriuresis in half the patients . It could be expected that an ANG II blocker would be better tolerated in cirrhotic patients, because bradykinin metabolism, and the production of NO and prostaglandins are not affected. Accordingly three recent studies have shown that low dose ANG II receptor type I blocking increased sodium excretion in cirrhotic patients without affecting systemic or renal hemodynamics, also in patients with normal systemic levels of renin-angiotensin-aldosterone. Losartan at a dose of 7.5 mg was able to counteract the sodium retention otherwise demonstrated in preascitic patients going from supine to standing position . Low dose Losartan could inhibit sodium retention when preascitic patients were given a high sodium diet . Losartan given at a higher dose -25 mg daily - to both preascitic and ascitic patients increased GFR and natriuresis without affection of blood pressure . In contrast to some previous results Schneider et al found that Losartan was able to reduce the portal pressure of cirrhotic patients at a dose at which the systemic circulation was not adversely affected, and even a natriuretic effect could be demonstrated . Accordingly a reducing effect of the ANG II antagonist Irbesartan has been demonstrated . Unfortunately an ameliorating effect of ANG II antagonists on portal pressure without adverse effects on blood pressure could not be demonstrated in two recent studies. A long-term (years) longitudinal study of cirrhotic patients with registration of consecutive changes in sodium handling, systemic and renal hemodynamics and neurohumoral regulations has never been done but is likely to elucidate the pathophysiology in these patients. In addition it is hypothesized that early intervention with the ANG II receptor antagonist Losartan could delay or even prevent development of the decompensated stage and thus improve survival and quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

The presence of cirrhosis in a liver biopsy; or, in the absence of histology, clinical and laboratory evidence of cirrhosis combined with years of excessive alcohol intake.

Age 18-70 years

Exclusion Criteria:

1. Cirrhosis due to alpha1-antitrypsin deficiency, viral hepatitis or autoimmunity.
2. Renal disease evidenced by proteinuria > 0,5 g/day.
3. Heart disease
4. Hypertension
5. Cancer or disease other than cirrhosis expected to limit life expectancy to < 5 years.
6. Pregnancy or lactation
7. Sepsis within 5 days
8. Gastrointestinal bleeding within 5 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2011-09

PRIMARY OUTCOMES:
Death

SECONDARY OUTCOMES:
varices
need for therapeutic ascites drainage
gastrointestinal bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Annette Dam, MD, Principal Investigator
Locations (1):
- Odense University Hospital, Odense, Odense, Denmark